CLINICAL TRIAL: NCT01927445
Title: Improving Stroke Prevention Therapy for Patients With Atrial Fibrillation in Primary Care: Protocol for a Pragmatic, Cluster-randomized Trial
Brief Title: Improving Stroke Prevention Therapy for Patients With Atrial Fibrillation in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: G-13-0001873
Record Dates: First submitted 2013-08-14; First posted 2013-08-22 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): No standardized intervention for management of patients with atrial fibrillation. Instead participants receive interventions for management of chronic kidney disease.
- quality improvement toolkit (Experimental): The toolkit includes provider-focused strategies (education, audit and feedback, electronic decision support and reminders) plus patient-directed strategies (educational letters and reminders).
  Interventions: Other: quality improvement toolkit

INTERVENTIONS:
Other: quality improvement toolkit — educational and informatics-based interventions, including brief guideline summary, decision support and audit and feedback
  Arms: quality improvement toolkit

SUMMARY:
The objective of this project is to increase the proportion of patients with AF that receive adequate stroke prevention therapy. Over half of patients with AF who suffer strokes are permanently disabled. Yet there remains a large portion of patients who do not receive appropriate stroke prevention therapy. The investigators hypothesize that a toolkit of quality improvement strategies in primary care could increase the proportion of patients with atrial fibrillation appropriately treated with stroke prevention therapy. The investigators' goal is to ensure the toolkit of interventions can be easily incorporated into day-to-day practice in primary care and can be readily and broadly disseminated if successful.

DETAILED DESCRIPTION:
The prevalence of atrial fibrillation (AF) is growing as the population ages and 15% of all strokes are already attributed to AF. Unfortunately, half of patients with AF do not receive prescriptions for anticoagulation to prevent stroke due to a variety of system, provider, and patient-level barriers. The investigators will conduct a pragmatic, cluster-randomized controlled trial to test a 'toolkit' of quality improvement interventions in primary care. In keeping with the recommendations of the chronic care model to simultaneously facilitate proactive care by providers and activate patients, the toolkit includes provider- focused strategies (education, audit and feedback, electronic medical record-based tools including decision support and reminders) plus patient-directed strategies (educational letters and reminders). Thirty three primary care clinics will be randomized to the intervention or usual care. The trial will last 12 months and will be powered to show a difference of 10% in the primary outcome of proportion of patients receiving guideline-concordant care for stroke prevention. Analysis will be blind to allocation.

ELIGIBILITY:
Inclusion Criteria:

* Physicians are participants in the Electronic Medical Record Administrative-data Linked Database (EMRALD).
* Patients are rostered to participating physicians, with a diagnosis in the chart of atrial fibrillation

Exclusion Criteria:

* Physicians who do not consent to data sharing
* Patients who change physicians during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2014-08; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with AF receiving guideline-concordant stroke prevention therapy | one year
  Patients with risk factors for stroke (ie. CHADS2 >1 or age >65) who are prescribed anticoagulants and patients with no risk factors for stroke (ie. CHADS2 = 0 and age <65) who are not prescribed anticoagulants will be considered to be receiving guideline concordant therapy. (For patients with CHADS2 = 1 but aged < 65 the guideline recommendations are unclear, so these patients will not be considered in the primary analysis. For example, in patients with AF and hypertension at a younger age, anticoagulation or aspirin or no treatment would each be reasonable.)

SECONDARY OUTCOMES:
proportion of patients taking warfarin in therapeutic range | one year
  patients must have INR measured 8 times during the year and therapeutic range assessed using Rosendaal method
proportion of patients taking a novel anticoagulant with appropriate dosing | one year
  Dabigatran, rivaroxaban and apixaban should be dose-adjusted in renal failure and avoided if estimated creatinine clearance is <30. Lower dose dabigatran is recommended for patients over 80.
proportion receiving aspirin | one year
proportion receiving clopidogrel | one year
proportion achieving target blood pressure | one year
  target defined as <130/80 for patients with diabetes, <150/80 for patients over 80, and <140/90 for all others

CONTACTS AND LOCATIONS:
Overall Officials: Karen Tu, MD, Principal Investigator — ICES
Locations (1):
- Institute for Clinical Evaluative Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee TM, Ivers NM, Bhatia S, Butt DA, Dorian P, Jaakkimainen L, Leblanc K, Legge D, Morra D, Valentinis A, Wing L, Young J, Tu K. Improving stroke prevention therapy for patients with atrial fibrillation in primary care: protocol for a pragmatic, cluster-randomized trial. Implement Sci. 2016 Dec 3;11(1):159. doi: 10.1186/s13012-016-0523-2. PMID 27912776